CLINICAL TRIAL: NCT02697201
Title: Dynamics of Muscle Mitochondria in Type 2 Diabetes (DYNAMMO-T2D)
Brief Title: Dynamics of Muscle Mitochondria in Type 2 Diabetes (DYNAMMO T2D)
Acronym: DYNAMMO-T2D
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Kirwan, Executive Director, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1311
Record Dates: First submitted 2016-02-18; First posted 2016-03-03 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Insulin Resistance
Keywords: Mitochondrial Dynamics; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — soybean oil, phospholipid emulsion; safflower oil, soybean oil, lecithin emulsion; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralipid Infusion, then Saline (Experimental): Participants in this arm will first receive a lipid infusion. Then 4 weeks later the saline infusion.
  Interventions: Drug: Intralipid; Drug: Saline
- Saline Infusion, then Intralipid (Sham Comparator): Participants in this arm will first receive a saline infusion. Then 4 weeks later the lipid infusion.
  Interventions: Drug: Intralipid; Drug: Saline

INTERVENTIONS:
Drug: Intralipid — 0.55 ml/kg/h
  Other Names: Liposyn
Drug: Saline — 0.55 ml/kg/h for

SUMMARY:
Insulin promotes the clearance of sugars from the blood into skeletal muscle and fat cells for use as energy; it also promotes storage of excess nutrients as fat. Type 2 diabetes occurs when the cells of the body become resistant to the effects of insulin, and this causes high blood sugar and contributes to a build-up of fat in muscle, pancreas, liver, and the heart. Understanding how insulin resistance occurs will pave the way for new therapies aimed at preventing and treating type 2 diabetes.

Mitochondria are cellular structures that are responsible for turning nutrients from food, into the energy that our cells run on. As a result, mitochondria are known as "the powerhouse of the cell." Mitochondria are dynamic organelles that can move within a cell to the areas where they are needed, and can fuse together to form large, string-like, tubular networks or divide into small spherical structures. The name of this process is "mitochondrial dynamics" and the process keeps the cells healthy. However, when more food is consumed compared to the amount of energy burned, mitochondria may become overloaded and dysfunctional resulting in a leak of partially metabolized nutrients that can interfere with the ability of insulin to communicate within the cell. This may be a way for the cells to prevent further uptake of nutrients until the current supply has been exhausted. However, long term overload of the mitochondria may cause blood sugar levels to rise and lead to the development of type 2 diabetes.

This study will provide information about the relationship between mitochondrial dynamics, insulin resistance and type 2 diabetes.

DETAILED DESCRIPTION:
The traditional view of mitochondria as isolated, spherical, energy producing organelles is undergoing a revolutionary transformation. Emerging data show that mitochondria form a dynamic networked reticulum that is regulated by cycles of fission and fusion. The discovery of a number of proteins that regulate these activities has led to important advances in understanding human disease. Data show that activation of dynamin related protein 1 (Drp1), a protein that controls mitochondrial fission, is reduced following exercise in prediabetes, and the decrease is linked to increased insulin sensitivity and fat oxidation. The proposed research will test the hypothesis that mitochondrial dynamics is a key mechanism of insulin resistance in type 2 diabetes. Translational first-in-man studies will use an acute lipid challenge to investigate the physiological significance of altered skeletal muscle mitochondrial dynamics on insulin sensitivity in humans. The experimental approach harnesses innovative molecular and cellular tools, interfaced with physiologically significant human studies to obtain meaningful data on insulin resistance, and has the potential to generate insights that will lead to new diabetes therapies for future generations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Sedentary
* Normal glucose tolerance
* BMI <25 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Effects of lipid infusion on mitochondrial fission | 5 years
  Fission will be assessed from quantitative measures of dynamin-related protein-1. The unit of assessment is arbitrary units of blot intensity and is expressed as AU.

SECONDARY OUTCOMES:
Effects of lipid infusion on mitochondrial function | 5 years
  Function will be assessed from oxygen consumption. Unit of assessment is pmol/s/mg of muscle.
Insulin sensitivity | 5 years
  Insulin sensitivity will be assessed by euglycemic hyperinsulinemic clamp. Units of assessment are mg/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: John P Kirwan, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Axelrod CL, Fealy CE, Erickson ML, Davuluri G, Fujioka H, Dantas WS, Huang E, Pergola K, Mey JT, King WT, Mulya A, Hsia D, Burguera B, Tandler B, Hoppel CL, Kirwan JP. Lipids activate skeletal muscle mitochondrial fission and quality control networks to induce insulin resistance in humans. Metabolism. 2021 Aug;121:154803. doi: 10.1016/j.metabol.2021.154803. Epub 2021 Jun 4. PMID 34090870